CLINICAL TRIAL: NCT04279639
Title: Observational Trial of Chaoyi Fanhuan Qigong as a Complementary Practice in Patients Receiving Treatment at a Tertiary-care Pain Management Unit: Part II
Brief Title: Observational Trial of Qigong for Patients in Pain
Status: Completed | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Mary Lynch, Principal Investigator, Nova Scotia Health Authority
Other Study IDs: 1021299
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Qigong

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- qigong practice: Patients in this arm participated in qigong as part of their treatment at the Pain Management Unit
  Interventions: Behavioral: qigong
- control: Patients attend the pain management unit but do not undertake qigong practice.

INTERVENTIONS:
Behavioral: qigong — Patients of the Pain Management Unit either experience usual treatment, or usual treatment plus qigong practice.
  Groups: qigong practice

SUMMARY:
This observational study documented outcomes resulting from qigong practice as a complementary self-care practice. All subjects continued with their usual medical care. Recruitment was passive, and participants consisted of those who encountered the practice as part of an earlier clinical trial, or entered the program prior to the observational period (posted information, word-of-mouth), or entered during the observational period (posted information).

ELIGIBILITY:
Inclusion Criteria:

* Those undertaking qigong practice as a complementary self-care practice at the Pain Management Unit

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the Pain Management Unit for management of chronic pain.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory | 8 week intervals
  Brief Pain Inventory, short form. Minimum is 0 (no pain), maximum is 10 (most pain)

SECONDARY OUTCOMES:
Profile of Mood States | 8 week intervals
  Profile of Mood States. Minimum is 30 (less depressed), maximum is 150 (more depressed)
health-related quality of life | 8 week intervals
  Short Form-12 item, Version 2 (SF-12V2). Minimum is 12 (lowest Quality of life), maximum is 56 (best Quality of life)
Sleep | 8 week intervals
  Pittsburg Sleep Quality Index. Minimum is 0 (best sleep), maximum is 21 (poor sleep).
Fatigue | 8 week intervals
  Chronic Fatigue Scale. Minimum is 0 (no fatigue), maximum is 42 (most fatigue).
Practice log | 8 week intervals
  Weekly Practice log

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Curry L, Pike M, Lynch M, Marcon D, Sawynok J. Observational Study of Qigong as a Complementary Self-Care Practice at a Tertiary-Care Pain Management Unit. Evid Based Complement Alternat Med. 2021 Jun 17;2021:6621069. doi: 10.1155/2021/6621069. eCollection 2021. PMID 34239585